CLINICAL TRIAL: NCT02032771
Title: Impact of M22 Synergistic Sequential Treatment (SST) Using Intense Pulsed Light and Fractional Non-ablative Photothermolysis on Skin Texture
Brief Title: Impact of M22 Synergistic Sequential Treatment (SST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-M22-IPL&ResurFX-13-02
Record Dates: First submitted 2014-01-06; First posted 2014-01-10 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Improvement of Wrinkles/Elastosis and/or Pigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- M22 IPL and ResurFX (Experimental): The procedure will include an intense pulse light (IPL) treatment followed by fractional non-ablative (FNA) treatment.
  Interventions: Device: M22 IPL and ResurFX

INTERVENTIONS:
Device: M22 IPL and ResurFX — The procedure will include an intense pulse light (M22 IPL) treatment followed by fractional non-ablative (M22 ResurFX) treatment.

SUMMARY:
Up to 40 healthy subjects at 2 sites, age 30-65 year old with Fitzpatrick-Elastosis score of 3-6 and mild to moderate age/sun-related facial pigmentation that wish to improve their facial skin appearance.

Hypothesis: The SST will improve the appearance of the wrinkles/elastosis and/or pigmentation by at least 1 on the FES scale or ≥50% in category scale at 3 months follow-ups in at least 50% of the study population.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and provide written Informed Consent;
2. Healthy adult, male or female, 30-65 years of age with Fitzpatrick-Goldman skin type I-V;
3. Having suitable facial areas with wrinkles Fitzpatrick-Goldman Wrinkle and Elastosis Score of 3-6 to be treated;
4. Having suitable facial areas with mild to moderate age/sun-related facial pigmentation
5. Able and willing to comply with the treatment/follow-up schedule and requirements;
6. Women of child-bearing age are required to be using a reliable method of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, Nova ring, partner with vasectomy or abstinence) at least 3 months prior to enrollment and throughout the course of the study.

Exclusion Criteria:

1. Skin type VI
2. Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 6 weeks after completion of breastfeeding
3. Heavy smoker (>1 pack of cigarettes a day)
4. Unable or unlikely to refrain from tanning, including the use of tanning booths, during the course of the study
5. Use of photosensitive medication for which light exposure is contraindicated.
6. Use of oral isotretinoin (Accutane®) within 3 months of initial treatment or during the course of the study. Note: skin must regain its normal degree of moisture prior to treatment.
7. Having indurate acne in treated area.
8. Any dermal/epidermal damage or disorder, mainly vascular or textural lesions, in treated area
9. Prior treatment, such as chemical peel (especially phenol based) or dermabrasion, in treated area within 3 months of initial treatment or during the course of the study;
10. Prior skin laser/light or another device treatment in treated area within 6 months of initial treatment or during the course of the study
11. Prior use of collagen, fat injections or other methods of skin augmentation (enhancement with injected or implanted material) in treated area within 12 months of initial treatment or during the course of the study. Treatment may not be performed at all over permanent dermal implants
12. Prior use of Botox in treatment area within 6 months
13. Prior ablative resurfacing procedure or face lift in treated area with laser or other devices within 12 months of initial treatment or during the course of the study
14. Any other surgery in treated area within 9 months of initial treatment or during the course of the study.
15. Participation in a study of another investigational device or drug involving the same anatomical site within 3 months prior to enrollment or during this evaluation, or if not involving the same anatomical site, as per the Investigator's discretion
16. History of keloid or any other type of hypertrophic scar formation or poor wound healing in a previously injured skin area
17. Showing symptoms of hormonal disorders, as per the Investigator's discretion (such as Melasma, Chloasma)
18. Concurrent inflammatory skin conditions, Open laceration or abrasion of any sort on area to be treated during the course of treatment
19. Active Herpes Simplex at the time of treatment or having experienced more than three episodes of Herpes Simplex eruption within a year of study enrollment;
20. Multiple dysplastic nevi in area to be treated
21. Having a bleeding disorder or taking anticoagulation medications, including heavy use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to treatment (as per the subject's physician discretion)
22. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications
23. Having any form of active cancer at the time of enrollment and during the course of the study or history of skin cancer on the face.
24. Pigmented lesion in the treated area that appears cancerous or is not deemed suitable for photo therapy, as determined by a dermatologist.
25. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the anesthesia, treatment, or healing process;
26. Mentally incompetent, prisoner or evidence of active substance or alcohol abuse
27. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study.
28. For subjects undergoing test spots: considerable undesired response consisting of skin hypopigmentation (long term whitening), a scar or pre scar formation, or any response deemed by the Investigator as grounds for exclusion.
29. Allergies to anesthetics.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with ≥ 50% improvement in Fitzpatrick Elastosis Scale (FES) | 3 months following 3rd treatment
  Skin improvement by Fitzpatrick Elastosis Scale (FES) or category scale at 3 months based on before/after photos

SECONDARY OUTCOMES:
Percentage of Participants with ≥ 50% improvement in Fitzpatrick Elastosis Scale (FES) | 1 and 6 months following 3rd treatment
  Overall skin improvement at 1 and 6 months by subject and investigator evaluation compared to baseline using the category global aesthetic improvement (GAI) scale
Change in erythema/ edema/ purpura and the response intensity | Following treatments- Baseline, 4, 8 weeks
  Immediate response (erythema, edema, purpura, etc.) of the skin will be assessed within 20-30 min post treatment by a 5 level scale: (0) None / (1) Trace / (2) Mild / (3) Moderate / (4) Severe.
Downtime in days | Following treatment- baseline, 4, 8 weeks
  Downtime defined as the period of time following the procedure during which the subject felt unable/unwilling to go out in public due to edema and / or erythema.
Subject Comfort using a Pain Visual Analogue Scale (VAS) | Following treatment- baseline, 4, 8 weeks
  Subject assessment of pain and discomfort associated with treatments using a Pain Visual Analogue Scale (VAS), were 0 is "no pain" and 100 is "intolerable pain".
Subject subjective assessment of improvement using categorical improvement scales | Following treatments- 4, 8 weeks and 1, 3 and 6 months follow up
  Subject subjective opinion of improvement and satisfaction with the treatment using the global aesthetic improvement (GAI) scale and pigment Improvement score.
Number of Participants with Adverse Events | Following treatment #1, 2 and 3 and all follow up visits
  Skin safety throughout the study as determined by the investigator by examining the post-treatment occurrences of complications and adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- Knight Dermatology Institute, Orlando, Florida, United States
- Konz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Knight JM, Kautz G. Sequential facial skin rejuvenation with intense pulsed light and non-ablative fractionated laser resurfacing in fitzpatrick skin type II-IV patients: A prospective multicenter analysis. Lasers Surg Med. 2019 Feb;51(2):141-149. doi: 10.1002/lsm.23007. Epub 2018 Aug 8. PMID 30091207